CLINICAL TRIAL: NCT07128134
Title: Evaluation of the Effects of the Low-level Laser Therapy as an Adjunct to Nonsurgical Treatment in Patients With Periimplantitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Aysegul SARI, Associate professor, Mustafa Kemal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KAEK-008-1/2025; 25.DHU.006 (Other Grant/Funding Number: Hatay Mustafa Kemal Univeristy Scientific Research Projects Commission)
Record Dates: First submitted 2025-07-31; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Periimplantitis
Keywords: Peri-implantitis; Laser therapy; Non-surgical treatment
MeSH Terms: conditions — Peri-Implantitis | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Laser treatment (Experimental): Laser Group: Group with peri-implantitis to receive low-level laser therapy in addition to non-surgical treatment of peri-implantitis)
  Interventions: Device: Low Level Laser Therapy; Procedure: Non-surgical Periodontal Treatment
- Non-surgical treatment (Active Comparator): Control group: Group with peri-implantitis who will undergo non-surgical treatment for peri-implantitis
  Interventions: Procedure: Non-surgical Periodontal Treatment

INTERVENTIONS:
Device: Low Level Laser Therapy — Although low-level laser therapy has been applied in cases of periodontitis, there are only a limited number of studies investigating its additional benefits in implants with peri-implantitis. This study aims to contribute to the literature on this subject.
  In addition to surgical periodontal treatment, low-level laser therapy (LLLT) was applied three times (on the same day as the initial treatment, on the third day, and on the seventh day) to the implants in the test group diagnosed with peri-implantitis. The 940 nm indium gallium arsenide phosphor diode laser (Epic Biolase, Irvine, CA, USA) will be applied perpendicular to the periodontal pocket for 20 seconds at a fixed distance of 15 mm and a continuous wavelength (3.41 J/cm2 application with a 1.76 cm2 spot and 0.3 W average output).
  Arms: Laser treatment
Procedure: Non-surgical Periodontal Treatment — Peri-implantitis diagnosis will be made in the control group, and non-surgical periodontal treatment of implants will be performed using titanium curettes (Hu-Friedy, Chicago, IL, USA).

SUMMARY:
The main objective of this study is to evaluate the clinical efficacy of low-level laser therapy (LLLT) in addition to non-surgical periodontal treatment in patients with peri-implantitis. The study aims to investigate the anti-inflammatory and regenerative effects of low-level laser therapy on peri-implant soft and hard tissues and to reveal its contribution to treatment success.

In this context, the specific objectives of the study are as follows:

1. To evaluate the effects of LLLT added to non-surgical mechanical treatment on clinical parameters such as plaque index, probing depth, bleeding index, and clinical attachment level.
2. To examine the contributions of laser therapy to tissue healing by analyzing biochemical markers in peri-implant sulcular fluid over time.

DETAILED DESCRIPTION:
This study will include volunteers who were diagnosed with peri-implantitis based on clinical and radiological examinations at the Department of Periodontology, Faculty of Dentistry, Hatay Mustafa Kemal University.

Seventy-two patients will be included in the study. In our study, patients will be divided into two groups. Thirty-six patients in the test group will receive low-level laser therapy in addition to non-surgical periodontal treatment. Thirty-six patients in the control group will receive only non-surgical periodontal treatment.

Periodontal indexes including plaque index, gingival index, bleeding on probing, probing pocket depth, and clinical attachment level will be recorded and peri-implant sulcus fluid will be collected from patients for routine diagnostic procedures. These measurements will be performed at baseline and at 1.5th and 3rd months by same researcher.

The following are required for a diagnosis of peri-implantitis:

1. Evidence of visual inflammatory changes in the soft tissues around the implant, accompanied by bleeding and/or suppuration during probing
2. Increased probing pocket depths compared to measurements obtained during the placement of the superstructure; and
3. Progressive bone loss according to radiographic bone level assessment within 1 year after delivery of the implant-supported prosthetic reconstruction; and
4. In cases where initial radiographs and probing depths are not available, a radiographic bone level of ≥3 mm and/or probing depths of ≥6 mm, along with the presence of bleeding, indicates peri-implantitis.

Study Treatment Protocol:

In the test group diagnosed with peri-implantitis, low-level laser therapy (LLLT) will be administered three times (on the same day as the initial treatment, on the 3rd day, and on the 7th day) in addition to non-surgical periodontal treatment by using A 940 nm indium gallium arsenide phosphor diode laser (Epic Biolase, Irvine, CA, USA).

PIOS regenerative (periostin) and inflammatory (vascular endothelial growth factor (VEGF), and interleukin-1 beta (IL-1ß)) biomarkers will be analyzed biochemically using the ELISA method (Enzyme-Linked Immunosorbent Assay) at the Department of Biochemistry, Faculty of Medicine, Hatay Mustafa Kemal University.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be willing to participate in the study.
* At least one implant with a pocket depth ≥ 6 mm and radiographic bone loss ≥ 3 mm diagnosed with peri-implantitis.
* Individuals aged 18-65.
* Patients who can understand and maintain oral hygiene education.

Exclusion Criteria:

* Individuals with any systemic disease that affects periodontal healing (diabetes, cancer, HIV/AIDS, acute infections, liver or kidney dysfunction/insufficiency, autoimmune disorders: rheumatoid arthritis, systemic lupus erythematosus, Hashimoto's thyroiditis)
* Female patients who are pregnant or breastfeeding
* Patients who have undergone periodontal treatment within the last six months
* Patients who have used antibiotics and regular anti-inflammatory medications within the last six months
* Use of medications that affect periodontal tissues (cyclosporine, phenytoin, sodium valproate, etc.).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in clinical peri-implant index values from baseline to the third months after non-surgical treatment with or without adjunctive low-level laser therapy | 0-3 month
  In peri-implantitis sites, Plaque Index (Silness-Löe), Gingival Index (Löe-Silness), bleeding on probing, probing pocket depth, and clinical attachment level scores will be recorded before and after non-surgical treatment with or without adjunctive low-level laser therapy

SECONDARY OUTCOMES:
Change from baseline to the third months after non-surgical treatment with or without adjunctive low-level laser therapy in the regenerative biomarker levels in patients with peri-implantitis | 0-3 month
  Periostin and vascular endothelial growth factor levels in peri-implant crevicular fluid will be measured before and after non-surgical treatment with or without adjunctive low-level laser therapy in peri-implantitis sites, using the ELISA immunoassay technique.

OTHER OUTCOMES:
Change from baseline to the third months after non-surgical treatment with or without adjunctive low-level laser therapy in the inflammatory biomarker levels in patients with peri-implantitis | 0-3 month
  Interleukin-1 beta levels in peri-implant crevicular fluid will be measured before and after non-surgical treatment with or without adjunctive low-level laser therapy in peri-implantitis sites, using the ELISA immunoassay technique.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet A Gunenc, DDs, Principal Investigator — Mustafa Kemal University; Aysegul Sari, PhD, Study Director — Mustafa Kemal University; Osman F Arpag, PhD, Study Chair — Mustafa Kemal University
Locations (1):
- Hatay Mustafa Kemal University, Hatay, Turkey (Türkiye)

REFERENCES:
- [Background] Gundogar H, Senyurt SZ, Erciyas K, Yalim M, Ustun K. The effect of low-level laser therapy on non-surgical periodontal treatment: a randomized controlled, single-blind, split-mouth clinical trial. Lasers Med Sci. 2016 Dec;31(9):1767-1773. doi: 10.1007/s10103-016-2047-z. Epub 2016 Aug 14. PMID 27523046
- [Background] Padial-Molina M, Volk SL, Taut AD, Giannobile WV, Rios HF. Periostin is down-regulated during periodontal inflammation. J Dent Res. 2012 Nov;91(11):1078-84. doi: 10.1177/0022034512459655. Epub 2012 Aug 29. PMID 22933606
- [Background] Santhosh VC, Karishma, Khader AA, Ramachandra V, Singh R, Shetty BK, Nimbalkar VK. Effect of periostin in peri-implant sulcular fluid and gingival crevicular fluid: A comparative study. Ann Afr Med. 2023 Oct-Dec;22(4):465-469. doi: 10.4103/aam.aam_171_22. PMID 38358147
- [Background] Barrientos S, Stojadinovic O, Golinko MS, Brem H, Tomic-Canic M. Growth factors and cytokines in wound healing. Wound Repair Regen. 2008 Sep-Oct;16(5):585-601. doi: 10.1111/j.1524-475X.2008.00410.x. PMID 19128254
- [Background] Aykol G, Baser U, Maden I, Kazak Z, Onan U, Tanrikulu-Kucuk S, Ademoglu E, Issever H, Yalcin F. The effect of low-level laser therapy as an adjunct to non-surgical periodontal treatment. J Periodontol. 2011 Mar;82(3):481-8. doi: 10.1902/jop.2010.100195. Epub 2010 Oct 8. PMID 20932157
- [Background] Saglam M, Kantarci A, Dundar N, Hakki SS. Clinical and biochemical effects of diode laser as an adjunct to nonsurgical treatment of chronic periodontitis: a randomized, controlled clinical trial. Lasers Med Sci. 2014 Jan;29(1):37-46. doi: 10.1007/s10103-012-1230-0. Epub 2012 Nov 16. PMID 23161345
- [Background] Carroll JD, Milward MR, Cooper PR, Hadis M, Palin WM. Developments in low level light therapy (LLLT) for dentistry. Dent Mater. 2014 May;30(5):465-75. doi: 10.1016/j.dental.2014.02.006. Epub 2014 Mar 21. PMID 24656472
- [Background] Karlsson MR, Diogo Lofgren CI, Jansson HM. The effect of laser therapy as an adjunct to non-surgical periodontal treatment in subjects with chronic periodontitis: a systematic review. J Periodontol. 2008 Nov;79(11):2021-8. doi: 10.1902/jop.2008.080197. PMID 18980508
- [Background] Wang CW, Renvert S, Wang HL. Nonsurgical Treatment of Periimplantitis. Implant Dent. 2019 Apr;28(2):155-160. doi: 10.1097/ID.0000000000000846. PMID 30913111
- [Background] Renvert S, Polyzois I, Claffey N. How do implant surface characteristics influence peri-implant disease? J Clin Periodontol. 2011 Mar;38 Suppl 11:214-22. doi: 10.1111/j.1600-051X.2010.01661.x. PMID 21323717
- [Background] Tomasi C, Wennstrom JL. Full-mouth treatment vs. the conventional staged approach for periodontal infection control. Periodontol 2000. 2009;51:45-62. doi: 10.1111/j.1600-0757.2009.00306.x. No abstract available. PMID 19878469
- [Background] Derks J, Schaller D, Hakansson J, Wennstrom JL, Tomasi C, Berglundh T. Effectiveness of Implant Therapy Analyzed in a Swedish Population: Prevalence of Peri-implantitis. J Dent Res. 2016 Jan;95(1):43-9. doi: 10.1177/0022034515608832. PMID 26701919
- [Background] Schwarz F, Derks J, Monje A, Wang HL. Peri-implantitis. J Periodontol. 2018 Jun;89 Suppl 1:S267-S290. doi: 10.1002/JPER.16-0350. PMID 29926957
- [Background] Berglundh T, Armitage G, Araujo MG, Avila-Ortiz G, Blanco J, Camargo PM, Chen S, Cochran D, Derks J, Figuero E, Hammerle CHF, Heitz-Mayfield LJA, Huynh-Ba G, Iacono V, Koo KT, Lambert F, McCauley L, Quirynen M, Renvert S, Salvi GE, Schwarz F, Tarnow D, Tomasi C, Wang HL, Zitzmann N. Peri-implant diseases and conditions: Consensus report of workgroup 4 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Clin Periodontol. 2018 Jun;45 Suppl 20:S286-S291. doi: 10.1111/jcpe.12957. PMID 29926491
- [Background] Schiegnitz E, Muller LK, Sagheb K, Theis L, Cagiran V, Kammerer PW, Wegener J, Wagner W, Al-Nawas B. Clinical long-term and patient-reported outcomes of dental implants in oral cancer patients. Int J Implant Dent. 2021 Jul 13;7(1):93. doi: 10.1186/s40729-021-00373-4. PMID 34255187